CLINICAL TRIAL: NCT03611335
Title: Effectiveness of the Consult for Addiction Treatment and Care in Hospitals (CATCH) Model for Engaging Patients in Opioid Use Disorder Treatment: Pragmatic Trial in a Large Municipal Hospital System
Brief Title: A Pragmatic Trial of the Consult for Addiction Treatment and Care in Hospitals (CATCH) Model for Engaging Patients in Opioid Use Disorder Treatment
Acronym: CATCH
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-00096
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Opioid Dependence; Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Site 1 H+H: Lincoln Medical and Mental Health Center
  Interventions: Behavioral: CATCH Interviews
- Site 2 H+H: Bellevue Hospital
  Interventions: Behavioral: CATCH Interviews
- Site 3 H+H: Metropolitan Hospital
  Interventions: Behavioral: CATCH Interviews
- Site 4 H+H: Elmhurst Hospital Center
  Interventions: Behavioral: CATCH Interviews
- Site 5 H+H: Coney Island Hospital
  Interventions: Behavioral: CATCH Interviews
- Site 6 H+H: Woodhull Medical and Mental Health Center
  Interventions: Behavioral: CATCH Interviews

INTERVENTIONS:
Behavioral: CATCH Interviews — Baseline interviews are conducted with CATCH staff (5/site); while Post-implementation interviews are conducted 9-12 months after introduction of CATCH, with CATCH staff (5/site) and patients (5/site)

SUMMARY:
This pragmatic clinical trial seeks to evaluate the effectiveness of the Consult for Addiction Treatment and Care in Hospitals (CATCH) intervention as a strategy for engaging patients with Opiod Use Disorder (OUD) in addiction treatment.

DETAILED DESCRIPTION:
The overarching objective of our study is to evaluate the effectiveness of CATCH as a strategy for engaging patients with OUD in MAT. A pragmatic trial at 6 hospitals, conducted in collaboration with the New York City Health and Hospitals system (H+H) and the New York City Department of Health and Mental Hygiene (DOHMH), will study the CATCH intervention in real-world settings and at scale. Guided by the RE-AIM evaluation framework, this hybrid effectiveness-implementation study (Type 1) focuses primarily on effectiveness, but also measures implementation outcomes to inform the intervention's adoption and sustainability. A rigorous stepped-wedge cluster randomized trial design determines the impact of CATCH on opioid treatment outcomes in comparison to usual care for a control period, followed by a 12-month intervention period and a maintenance period, and utilizes existing administrative data to evaluate outcomes. Aim 1 (primary aim) is to evaluate the effectiveness of CATCH in increasing post-discharge initiation and engagement in MAT, defined respectively as receiving outpatient MAT within 14 days of discharge, and having at least 2 additional MAT visits in the first month. Aim 2 is to assess the effectiveness of CATCH for increasing treatment retention, defined as continuous receipt of MAT for 6 months. Aim 3 is to compare the frequency of acute care utilization and overdose deaths, and their associated costs, among patients with OUD who are hospitalized during the CATCH period versus usual care. Aim 4 is to evaluate implementation outcomes at CATCH sites using a mixed methods approach to assess the intervention's Reach (proportion of eligible patients reached); Adoption (utilization by medical staff); and Implementation fidelity (barriers to delivering high-quality MAT).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years);
* Hospitalized for at least 1 night on an inpatient service (not including intensive care);
* Admission or discharge diagnosis (based on ICD-10 codes) of opioid use disorder or opioid poisoning.

Cases are excluded if they received MAT (buprenorphine, methadone maintenance treatment, or naltrexone) in the 30 days prior to admission. Cases included in the intervention condition must have been admitted on a date following implementation of CATCH.

Exclusion Criteria:

* Lack of fluency in English, unable to provide informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study retrospectively analyzes administrative data for patients with OUD who have been hospitalized at the participating sites. These patients are not recruited or enrolled.The cases identified through administrative data consists of individuals with OUD who are hospitalized at one of the six study sites. We anticipate that the characteristics of this population will vary by site, given the differences in patient populations served by each of the participating hospitals. Overall, we expect that cases will have the following demographic characteristics: 28% female; 14% Hispanic; 24% Black, 37% White, 1% Asian, 38% mixed race/other; 4% age 18-25, 33% age 26-45, 55% age 46-65, 7% >65 years.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Effectiveness of CATCH in increasing MAT initiation among patients with OUD. | Initiate MAT outpatient treatment within 14 days of discharge.
  Effectiveness of patients hospitalized during the CATCH period to have higher rates of treatment initiation.
Effectiveness of CATCH in increasing MAT engagement among patients with OUD. | Have 2 or more additional MAT services within 30 days of treatment initiation.
  Effectiveness of patients hospitalized during the CATCH period to have higher rates of treatment engagement, defined as having 2 or more additional MAT services within 30 days of treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNeely, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The individual patient data collected for this study will not be made available to others, as data has been extracted from New York State Medicaid claims, which is highly confidential. The data use agreement which allows the study team access to this data does not permit sharing with individuals unless they are approved by New York State.

REFERENCES:
- [Derived] Rostam-Abadi Y, Wang S, King C, Kalyanaraman Marcello R, Van Wye G, Tuazon E, Kennedy J, Cooke C, Mazumdar M, Tarpey T, Billings J, Appleton N, Fernando J, Fawole A, Siddiqui S, Barron C, Schatz D, McNeely J. Addiction Consult Services, Mortality, and Acute Care Utilization in Inpatients With Opioid Use Disorder: A Secondary Analysis of a Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2525222. doi: 10.1001/jamanetworkopen.2025.25222. PMID 40768148
- [Derived] McNeely J, Wang SS, Rostam Abadi Y, Barron C, Billings J, Tarpey T, Fernando J, Appleton N, Fawole A, Mazumdar M, Weinstein ZM, Kalyanaraman Marcello R, Dolle J, Cooke C, Siddiqui S, King C. Addiction Consultation Services for Opioid Use Disorder Treatment Initiation and Engagement: A Randomized Clinical Trial. JAMA Intern Med. 2024 Sep 1;184(9):1106-1115. doi: 10.1001/jamainternmed.2024.3422. PMID 39073796
- [Derived] McNeely J, Troxel AB, Kunins HV, Shelley D, Lee JD, Walley A, Weinstein ZM, Billings J, Davis NJ, Marcello RK, Schackman BR, Barron C, Bergmann L. Study protocol for a pragmatic trial of the Consult for Addiction Treatment and Care in Hospitals (CATCH) model for engaging patients in opioid use disorder treatment. Addict Sci Clin Pract. 2019 Feb 19;14(1):5. doi: 10.1186/s13722-019-0135-7. PMID 30777122